CLINICAL TRIAL: NCT03510143
Title: Effect of Polyglycolic Acid Mesh (Neoveil) for Reducing Drain Amount and Chyle Leakage After Thyroid Cancer Surgery: A Prospective, Randomized Controlled Study
Brief Title: Effect of Polyglycolic Acid Mesh (Neoveil) in Thyroid Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Green Cross Corporation (Industry)
Responsible Party: Principal Investigator, Jin Wook Yi, Clinical Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1802-087-923
Record Dates: First submitted 2018-03-20; First posted 2018-04-27 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Thyroid Gland Carcinoma; Thyroid Cancer; Thoracic Duct Leak
Keywords: thyroid cancer; Neoveil; seroma; chyle leakage
MeSH Terms: conditions — Thyroid Neoplasms; Seroma

STUDY DESIGN:
Intervention Model Description: Neoveil applied // Neoveil non-applied
Who Masked: Participant
Masking Description: Participants cannot know the Neoveil apply in their surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No use of Neoveil in the neck node dissection area
- Neoveil (Experimental): Use of Neoveil in the neck node dissection area
  Interventions: Device: Neoveil (Polyglycolic Acid Mesh)

INTERVENTIONS:
Device: Neoveil (Polyglycolic Acid Mesh) — Apply the Neoveil (Polyglycolic Acid Mesh) in the neck node dissection area in thyroid cancer surgery.
  Arms: Neoveil

SUMMARY:
This study is a randomized controlled study to investigate the effect of "Polyglycolic Acid Mesh Sheet (NeoveilTM)" on the thyroid cancer surgery.

DETAILED DESCRIPTION:
Thyroid cancer is a most common solid organ cancer in South Korea, according to 2014 statistics from Korea Central Cancer Registry.

The most important treatment of thyroid cancer is a surgery. Principle of thyroid cancer surgery is cancer-involved thyroid gland resection and central/lateral compartment of neck node dissection.

Part of surgical complications associated with neck lymph node dissection are seroma and chyle leakage. Incidence of seroma and chyle leakage have been reported as 4-5% and 1-7% in previous studies. Currently, there's no effective agents to prevent these complications.

"Polyglycolic Acid Mesh Sheet (NeoveilTM)" is a tissue strengthening repair agent which is prevent air or fluid leakage. It's effects were proven in various surgical field - prevent air leakage in lung surgery, reduce pancreatic fistula in pancreas surgery and so on. However, there's no result in thyroid cancer surgery.

This study will investigate the usability of NeoveilTM in thyroid cancer surgery and have the effect of preventing seroma and chyle leakage.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are between 20 and 70 years of age
* Patients who agreed to the study
* Patients undergoing thyroidectomy and cervical node dissection for thyroid cancer
* Patients without perithyroidal organ infiltration or distant metastasis
* Before the operation, bilateral vocal cord movement was normal
* Patients without significant abnormal findings in laboratory tests before surgery

Exclusion Criteria:

* Patients judged to be inadequate by the person in charge of clinical trial
* Aspirin, anti-platelet medication within 7 days of admission
* Uncontrolled hypertension, diabetes, chronic renal failure, coagulation disorders
* Cardiovascular disease (angina, heart failure, myocardial infarction, history of coronary artery disease, stroke, transient ischemic attack)
* Drug abuse and alcohol abuse
* History of esophagus and airway diseases
* Patients who participated in other clinical trials within 30 days
* Patients who had previous history of neck irradiation or neck surgery
* Patients with a history of allergy to drugs
* For women, pregnant and lactating patients

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of triglyceride(TG) level in drained fluid | Change from drain TG level from postoperative 1st day to postoperative 2nd day
  Triglyceride level in the drained fluid, check time 9:00AM, unit : mg/dL

SECONDARY OUTCOMES:
Drain amount | Postoperative 1st and 2nd days
  Drained fluid amount during 24 hours (Baseline 6:00 AM), unit : ml

CONTACTS AND LOCATIONS:
Locations (1):
- Jin Wook Yi, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jang JY, Shin YC, Han Y, Park JS, Han HS, Hwang HK, Yoon DS, Kim JK, Yoon YS, Hwang DW, Kang CM, Lee WJ, Heo JS, Kang MJ, Chang YR, Chang J, Jung W, Kim SW. Effect of Polyglycolic Acid Mesh for Prevention of Pancreatic Fistula Following Distal Pancreatectomy: A Randomized Clinical Trial. JAMA Surg. 2017 Feb 1;152(2):150-155. doi: 10.1001/jamasurg.2016.3644. PMID 27784046
- [Result] Kuwata T, Shinohara S, Takenaka M, Oka S, Chikaishi Y, Hirai A, Kuroda K, So T, Tanaka F. The impact of covering the bulla with an absorbable polyglycolic acid (PGA) sheet during pneumothorax surgery. Gen Thorac Cardiovasc Surg. 2016 Sep;64(9):558-60. doi: 10.1007/s11748-015-0545-8. Epub 2015 Apr 10. PMID 25860987
- [Result] Kobayashi S, Takeda Y, Nakahira S, Tsujie M, Shimizu J, Miyamoto A, Eguchi H, Nagano H, Doki Y, Mori M. Fibrin Sealant with Polyglycolic Acid Felt vs Fibrinogen-Based Collagen Fleece at the Liver Cut Surface for Prevention of Postoperative Bile Leakage and Hemorrhage: A Prospective, Randomized, Controlled Study. J Am Coll Surg. 2016 Jan;222(1):59-64. doi: 10.1016/j.jamcollsurg.2015.10.006. Epub 2015 Oct 23. PMID 26597705